CLINICAL TRIAL: NCT02669108
Title: PET-MRI for Functional Imaging of the Testis: A New Methodology for Evaluation of the Infertile Male
Brief Title: PET-MRI for Functional Imaging of the Testis: A Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-01636
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Infertility; Non-obstructive Azoospermia; Vasectomy
Keywords: testis; spermatogenesis
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PET/MRI of the Testis (Other): PET/MRI of the testis will be performed upon the patient achieving azoospermia (following the vasectomy), or 25 ejaculations and following proven azoospermia (via standard of care semen analysis).
  Interventions: Device: PET/ MRI of the Testis

INTERVENTIONS:
Device: PET/ MRI of the Testis — PET/MRI of the testis will be performed upon the patient achieving azoospermia (following the vasectomy), or 25 ejaculations and following proven azoospermia (via standard of care semen analysis).

SUMMARY:
The primary objective of this study is to explore feasibility of testis functionality assessment and testis imaging obtained from Positron Emissions Tomography (PET) /Magnetic Resonance Imagine (MRI). Using advanced MRI metrics, investigators will study the three-dimensional structure of normal testis, the levels of specific elements and compounds in the tissues (which can only be found via these imaging techniques), and the directionality (and alterations in directionality) of tissue structure. Investigators hope to develop hypothesis that will in turn suggest bio-markers to be explored in subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Men with proven paternity desiring vasectomy who are over 18 years of age.

Exclusion Criteria:

* Bilaterally absent testes, unilaterally or bilaterally undescended testes
* Patients who have proven azoospermia or no proven paternity
* Inability to tolerate MRI including conditions such as claustrophobia or inability to lay flat for > 45 minutes.
* Presence of pacemaker/IImplantable Cardioverter Defibrillator (ICD) or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants.
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study
* All women are excluded as such patients do not have the relevant anatomy being considered in this study
* Anyone from a vulnerable population will be excluded from the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Diffusion-weighted coefficient imaging of testis using PET/MRI fusion | 2 Months
T2 relaxation time using PET/MRI fusion | 2 Months
Metabolite concentration using PET/MRI fusion | 2 Months
Spectroscopy of the testis using PET/MRI fusion | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Alukal, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States